CLINICAL TRIAL: NCT03073720
Title: Correlation Between Follicular Fluid Levels of Bioavailable Vitamin D and Embryo Quality Markers: Euploid Status, Morphokinetics and Mitochondrial DNA Content Among UAE Women Undergoing an IVF Cycle
Brief Title: Follicular Fluid, Bioavailable Vitamin D and Embryo Quality Markers
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Prof Dr. Human Fatemi, Medical Director, ART Fertility Clinics LLC
Other Study IDs: 1606-ABU-048-HF
Record Dates: First submitted 2017-02-27; First posted 2017-03-08 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — follicular fluid,serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the correlation between bioavailable Vitamin D values and euploid status of the embryos in larger size follicles from UAE women undergoing in vitro fertilization procedures.

DETAILED DESCRIPTION:
To study the possible correlation between bioavailable vitamin D values in follicular fluid and embryo quality markers.

To correlate bioavailable Vitamin D values in follicular fluid from large size follicles with embryo euploid status as our main objective. Secondly, looking at morphokinetics and mitochondrial content of these embryos.

Taking into account that most of UAE patients have deficiency or insufficiency of Vitamin D, if there is a correlation found we will understand better the underlying mechanism by which bioavailable Vitamin D levels may be affecting embryo quality, therefore IVF outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women´s Age >18 - ≤43 years.
* BMI 19-33
* Male partner will produce fresh sperm sample on the same day of the egg collection procedure.
* Women with more than 10 follicles at the time of the trigger
* At the time of egg retrieval, at least three follicles between 14-<17 mm and three follicles ≥17 mm.
* Women ≤35 years old stimulation with rFSH antagonist
* Women ≥36 years old stimulation with highly-purified human menopausal gonadotropins (hpHMG) specifically for the additional LH.
* Middle East population

Exclusion Criteria:

* Polycystic ovarian syndrome (according to the Rotterdam Criteria).
* Patients at risk of OHSS, according to the criteria previously described by Papanikolau et al. (23).
* History of endometriosis, classified according to the American Fertility Society (AFS) as stage 3 or more.
* Severe male factor definition (<2 million of sperm per ml of ejaculate)
* Recurrent miscarriage (3 miscarriages)
* Smokers
* History of chemotherapy or radiotherapy

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: UAE patients with infertility (primary or secondary) and indication for IVF/ICSI treatment with PGS
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D values in follicular fluid and embryo quality markers among UAE women undergoing an IVF cycle | 6-10 months
  A correlation between vitamin D levels and embryo development patterns

CONTACTS AND LOCATIONS:
Overall Officials: Human Fatemi, Medical D., Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Grober U, Spitz J, Reichrath J, Kisters K, Holick MF. Vitamin D: Update 2013: From rickets prophylaxis to general preventive healthcare. Dermatoendocrinol. 2013 Jun 1;5(3):331-47. doi: 10.4161/derm.26738. Epub 2013 Nov 5. PMID 24516687
- [Background] Anagnostis P, Karras S, Goulis DG. Vitamin D in human reproduction: a narrative review. Int J Clin Pract. 2013 Mar;67(3):225-35. doi: 10.1111/ijcp.12031. Epub 2013 Jan 7. PMID 23294318
- [Background] Coney P, Demers LM, Dodson WC, Kunselman AR, Ladson G, Legro RS. Determination of vitamin D in relation to body mass index and race in a defined population of black and white women. Int J Gynaecol Obstet. 2012 Oct;119(1):21-5. doi: 10.1016/j.ijgo.2012.05.024. Epub 2012 Jul 18. PMID 22818533
- [Background] Irani M, Minkoff H, Seifer DB, Merhi Z. Vitamin D increases serum levels of the soluble receptor for advanced glycation end products in women with PCOS. J Clin Endocrinol Metab. 2014 May;99(5):E886-90. doi: 10.1210/jc.2013-4374. Epub 2014 Feb 27. PMID 24606102
- [Background] Hussain AN, Alkhenizan AH, El Shaker M, Raef H, Gabr A. Increasing trends and significance of hypovitaminosis D: a population-based study in the Kingdom of Saudi Arabia. Arch Osteoporos. 2014;9:190. doi: 10.1007/s11657-014-0190-3. Epub 2014 Sep 12. PMID 25213798
- [Background] Farzadi L, Khayatzadeh Bidgoli H, Ghojazadeh M, Bahrami Z, Fattahi A, Latifi Z, Shahnazi V, Nouri M. Correlation between follicular fluid 25-OH vitamin D and assisted reproductive outcomes. Iran J Reprod Med. 2015 Jun;13(6):361-6. PMID 26330851
- [Background] Parikh G, Varadinova M, Suwandhi P, Araki T, Rosenwaks Z, Poretsky L, Seto-Young D. Vitamin D regulates steroidogenesis and insulin-like growth factor binding protein-1 (IGFBP-1) production in human ovarian cells. Horm Metab Res. 2010 Sep;42(10):754-7. doi: 10.1055/s-0030-1262837. Epub 2010 Aug 13. PMID 20711952
- [Background] Ozkan S, Jindal S, Greenseid K, Shu J, Zeitlian G, Hickmon C, Pal L. Replete vitamin D stores predict reproductive success following in vitro fertilization. Fertil Steril. 2010 Sep;94(4):1314-1319. doi: 10.1016/j.fertnstert.2009.05.019. Epub 2009 Jul 8. PMID 19589516
- [Background] Anifandis GM, Dafopoulos K, Messini CI, Chalvatzas N, Liakos N, Pournaras S, Messinis IE. Prognostic value of follicular fluid 25-OH vitamin D and glucose levels in the IVF outcome. Reprod Biol Endocrinol. 2010 Jul 28;8:91. doi: 10.1186/1477-7827-8-91. PMID 20667111
- [Background] Rudick B, Ingles S, Chung K, Stanczyk F, Paulson R, Bendikson K. Characterizing the influence of vitamin D levels on IVF outcomes. Hum Reprod. 2012 Nov;27(11):3321-7. doi: 10.1093/humrep/des280. Epub 2012 Aug 21. PMID 22914766
- [Background] Franasiak JM, Molinaro TA, Dubell EK, Scott KL, Ruiz AR, Forman EJ, Werner MD, Hong KH, Scott RT Jr. Vitamin D levels do not affect IVF outcomes following the transfer of euploid blastocysts. Am J Obstet Gynecol. 2015 Mar;212(3):315.e1-6. doi: 10.1016/j.ajog.2014.09.029. Epub 2014 Oct 11. PMID 25265402
- [Background] Bikle DD, Gee E, Halloran B, Kowalski MA, Ryzen E, Haddad JG. Assessment of the free fraction of 25-hydroxyvitamin D in serum and its regulation by albumin and the vitamin D-binding protein. J Clin Endocrinol Metab. 1986 Oct;63(4):954-9. doi: 10.1210/jcem-63-4-954. PMID 3745408
- [Background] Powe CE, Evans MK, Wenger J, Zonderman AB, Berg AH, Nalls M, Tamez H, Zhang D, Bhan I, Karumanchi SA, Powe NR, Thadhani R. Vitamin D-binding protein and vitamin D status of black Americans and white Americans. N Engl J Med. 2013 Nov 21;369(21):1991-2000. doi: 10.1056/NEJMoa1306357. PMID 24256378
- [Background] Engelman CD, Fingerlin TE, Langefeld CD, Hicks PJ, Rich SS, Wagenknecht LE, Bowden DW, Norris JM. Genetic and environmental determinants of 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D levels in Hispanic and African Americans. J Clin Endocrinol Metab. 2008 Sep;93(9):3381-8. doi: 10.1210/jc.2007-2702. Epub 2008 Jul 1. PMID 18593774
- [Background] Diez-Juan A, Rubio C, Marin C, Martinez S, Al-Asmar N, Riboldi M, Diaz-Gimeno P, Valbuena D, Simon C. Mitochondrial DNA content as a viability score in human euploid embryos: less is better. Fertil Steril. 2015 Sep;104(3):534-41.e1. doi: 10.1016/j.fertnstert.2015.05.022. Epub 2015 Jun 11. PMID 26051102
- [Background] Seli E. Mitochondrial DNA as a biomarker for in-vitro fertilization outcome. Curr Opin Obstet Gynecol. 2016 Jun;28(3):158-63. doi: 10.1097/GCO.0000000000000274. PMID 27077472
- [Background] Fragouli E, Spath K, Alfarawati S, Kaper F, Craig A, Michel CE, Kokocinski F, Cohen J, Munne S, Wells D. Altered levels of mitochondrial DNA are associated with female age, aneuploidy, and provide an independent measure of embryonic implantation potential. PLoS Genet. 2015 Jun 3;11(6):e1005241. doi: 10.1371/journal.pgen.1005241. eCollection 2015 Jun. PMID 26039092
- [Background] Blomberg Jensen M. Vitamin D and male reproduction. Nat Rev Endocrinol. 2014 Mar;10(3):175-86. doi: 10.1038/nrendo.2013.262. Epub 2014 Jan 14. PMID 24419359
- [Background] Saadi HF, Nagelkerke N, Benedict S, Qazaq HS, Zilahi E, Mohamadiyeh MK, Al-Suhaili AI. Predictors and relationships of serum 25 hydroxyvitamin D concentration with bone turnover markers, bone mineral density, and vitamin D receptor genotype in Emirati women. Bone. 2006 Nov;39(5):1136-1143. doi: 10.1016/j.bone.2006.05.010. Epub 2006 Jun 30. PMID 16814623
- [Background] Aleyasin A, Hosseini MA, Mahdavi A, Safdarian L, Fallahi P, Mohajeri MR, Abbasi M, Esfahani F. Predictive value of the level of vitamin D in follicular fluid on the outcome of assisted reproductive technology. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):132-7. doi: 10.1016/j.ejogrb.2011.07.006. Epub 2011 Aug 10. PMID 21835540
- [Background] Yousefzadeh P, Shapses SA, Wang X. Vitamin D Binding Protein Impact on 25-Hydroxyvitamin D Levels under Different Physiologic and Pathologic Conditions. Int J Endocrinol. 2014;2014:981581. doi: 10.1155/2014/981581. Epub 2014 Apr 28. PMID 24868205
- [Background] Papanikolaou EG, Humaidan P, Polyzos N, Kalantaridou S, Kol S, Benadiva C, Tournaye H, Tarlatzis B. New algorithm for OHSS prevention. Reprod Biol Endocrinol. 2011 Nov 3;9:147. doi: 10.1186/1477-7827-9-147. PMID 22054506
- [Background] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Background] Van Steirteghem AC, Nagy Z, Joris H, Liu J, Staessen C, Smitz J, Wisanto A, Devroey P. High fertilization and implantation rates after intracytoplasmic sperm injection. Hum Reprod. 1993 Jul;8(7):1061-6. doi: 10.1093/oxfordjournals.humrep.a138192. PMID 8408487
- [Background] Devroey P, Liu J, Nagy Z, Goossens A, Tournaye H, Camus M, Van Steirteghem A, Silber S. Pregnancies after testicular sperm extraction and intracytoplasmic sperm injection in non-obstructive azoospermia. Hum Reprod. 1995 Jun;10(6):1457-60. doi: 10.1093/humrep/10.6.1457. PMID 7593514
- [Background] Van Landuyt L, De Vos A, Joris H, Verheyen G, Devroey P, Van Steirteghem A. Blastocyst formation in in vitro fertilization versus intracytoplasmic sperm injection cycles: influence of the fertilization procedure. Fertil Steril. 2005 May;83(5):1397-403. doi: 10.1016/j.fertnstert.2004.10.054. PMID 15866575
- [Background] Staessen C, Platteau P, Van Assche E, Michiels A, Tournaye H, Camus M, Devroey P, Liebaers I, Van Steirteghem A. Comparison of blastocyst transfer with or without preimplantation genetic diagnosis for aneuploidy screening in couples with advanced maternal age: a prospective randomized controlled trial. Hum Reprod. 2004 Dec;19(12):2849-58. doi: 10.1093/humrep/deh536. Epub 2004 Oct 7. PMID 15471934
- [Background] Scott RT, Hofmann GE, Muasher SJ, Acosta AA, Kreiner DK, Rosenwaks Z. Correlation of follicular diameter with oocyte recovery and maturity at the time of transvaginal follicular aspiration. J In Vitro Fert Embryo Transf. 1989 Apr;6(2):73-5. doi: 10.1007/BF01130729. PMID 2723509
- [Background] Alikani M, Calderon G, Tomkin G, Garrisi J, Kokot M, Cohen J. Cleavage anomalies in early human embryos and survival after prolonged culture in-vitro. Hum Reprod. 2000 Dec;15(12):2634-43. doi: 10.1093/humrep/15.12.2634. PMID 11098037
- [Background] Vermeulen A, Verdonck L, Kaufman JM. A critical evaluation of simple methods for the estimation of free testosterone in serum. J Clin Endocrinol Metab. 1999 Oct;84(10):3666-72. doi: 10.1210/jcem.84.10.6079. PMID 10523012
- [Background] Meseguer M, Herrero J, Tejera A, Hilligsoe KM, Ramsing NB, Remohi J. The use of morphokinetics as a predictor of embryo implantation. Hum Reprod. 2011 Oct;26(10):2658-71. doi: 10.1093/humrep/der256. Epub 2011 Aug 9. PMID 21828117